CLINICAL TRIAL: NCT04001257
Title: Role of 18F-Fluoro-Ethyl-Tyrosine (FET) Positron Emission Tomography (PET) for Grading Glioma
Brief Title: 18F-Fluoro-Ethyl-Tyrosine (FET) Positron Emission Tomography (PET) and Grading Glioma
Acronym: GLIOFET
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: GLIOFET (29BRC19.0140)
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Positron Emission Tomography; Glioma
Keywords: 18F-FET PET; glioma; grading
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Role of 18F-FET PET for grading gliomas according to 2016 WHO classification: value of quantitative and qualitative data obtained by 18F-FET PET for differentiating low grade glioma (WHO II) versus high grade gliomas (WHO III and IV)

DETAILED DESCRIPTION:
The management and prognosis of patients with glioma is highly dependent on the tumour grade according to the new 2016 classification of the World Health Organization (WHO), which incorporates molecular characteristics. Standard magnetic resonance imaging (MRI) enhanced by contrast is the basis of imaging primary brain tumours including gliomas. Nevertheless MRI specificity to type glioma is limited. Recently, positron emission tomography (PET) molecular imaging using radiolabeled amino acids or their analogues has been recommended by the Neuro-Oncology Response Assessment (RANO) working group for differential diagnosis of brain lesions, non-invasive classification of glial tumours, prognostic value, tumour delineation, stereotactic biopsy radiotherapy planification and treatments follow-up, to provide additional informations beyond MRI on biological processes such as cell proliferation, membrane biosynthesis, glucose consumption and absorption of amino acid analogues. Among the radiotracers used in PET, radiolabeled amino acids or their analogues are increasingly used in clinical routine for glioma imaging. Although most previous PET studies focused on brain gliomas used L-[methyl- 11 C] -methionine (11C-MET), the fluorinated amino acid analogue O - (2-[ 18 F] fluoroethyl) -L-tyrosine (18F-FET) appeared to be a favorable marker for clinical routine due to his longer half-life than Carbone 11. Recent european guidelines attempt to provide some guidance on the performance and interpretation of molecular imaging. The authors recommend a static (20-40 mn after injection (Pi)) or dynamic PET acquisition (40-50 mn from injection). A visual analysis can be completed by a quantitative analysis which consists to measure mean and maximal tumour activity uptake values (SUVmean and SUVmax) and their respective tumour to background ratios (TBRmean and TBRmax). Although the mean physiological brain activity uptake is well defined, the measurement of mean glioma activity uptake is less clear. Indeed, TBRmean depends on the delineation of the tumour ROI and/or VOI. Most often previously, VOI was determined by a 3D contouring process using a tumour-to-brain ratio of at least 1.6 at the beginning of the scan, threshold defined on a brain gliomas biopsy-controlled study. Moreover, Albert et al. emphasized the interest of early TBRmax.To our knowledge, none study evaluated others parameters as SUVmax, SUVmean and TBRmean in early period. In this context, the aim of this study was to compare quantitative and qualitative PET parameters between Low Grade Glioma and High Grade Glioma.

ELIGIBILITY:
Inclusion Criteria:

* glial tumor
* patient underwent 18F-FET PET at Brest University Hospital
* no opposite to participate

Exclusion Criteria:

* patient Under 18 years old
* opposite to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with glioma histologically proven (grades II, III and IV according to WHO 2016) underwent 18F-FET PET at Brest university hospital
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
quantitative criteria (SUVmax) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study mean value of SUVmax obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)
quantitative criteria (TBRmax) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study mean value of TBRmax obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)
quantitative criteria (SUVmean) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study mean value of SUVmean obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)
quantitative criteria (TBRmean) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study mean value of TBRmean obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)
quantitative criteria (SUVpeak) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study mean value of SUVpeak obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)
quantitative criteria (métabolic tumoral volume MTV) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study mean value of MTV obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)
quantitative criteria (Total Lesion Glycolysis TLG) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study mean value of TLG obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)
quantitative criteria (SUVmin) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study mean value of SUVmin obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)

SECONDARY OUTCOMES:
qualitative criteria (Time Activity Curve TAC) between 2 groups (glioma II vs glioma III-IV) | 3 months
  study qualitative data obtained by 18F-FET PET between 2 groups (glioma II vs glioma III-IV)
agreement between readers for quantitative and qualitative criteria | 3 months
  study inter and intra observers agreement
diagnostic accuracy of clinical data to discriminate the 2 groups of glioma (symptom or size of tumor) | 3 months
  study diagnostic accuracy of clinical data
diagnostic accuracy of biological criteria (as MGMT mutation or IDH status or 1p19q codeletion, ATRX status) to discriminate the 2 groups of glioma | 3 months
  study diagnostic accuracy of biological data
diagnostic accuracy of PET criteria (SUVmax, TBRmax, SUVmean, TBRmean, SUVpeak, SUVmin, TLG and MTV) between the 2 groups of glioma | 3 months
  study diagnostic accuracy of PET data
prognostic value of F-FET PET data on PET Baseline on PFS | 2 years and 3 months
  study the prognostic value of PET criteria on PFS
prognostic value of F-FET PET data on PET Baseline on OS | 2 years and 3 months
  study the prognostic value of PET criteria on OS
prognostic value of variation of quantitative PET data (SUVmax, TBRmax, SUVmean, TBRmean, SUVpeak, SUVmin, MTV, TLG) (for example deltaSUVmax between PET Baseline and PET 3 months) on PFS | 2 years and 3 months
  modification of PET criteria between PET Baseline and PET at follow-up and their prognostic value on PFS
prognostic value of variation of quantitative PET data (SUVmax, TBRmax, SUVmean, TBRmean, SUVpeak, SUVmin, MTV, TLG) (for example deltaSUVmax between PET Baseline and PET 3 months) on OS | 2 years and 3 months
  modification of PET criteria between PET Baseline and PET at follow-up and their prognostic value on OS

CONTACTS AND LOCATIONS:
Overall Officials: solene querellou, MD, Study Chair — CHRU Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning Two and ending fivethree years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.